CLINICAL TRIAL: NCT01197313
Title: Depression and Quality of Life in Chronic Heart Failure Patients and the Caregivers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Ying-Tai Wu/ Associate professor, School and Graduate Institute of Physical Therapy, College of Medicine, National Taiwan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 9561709097
Record Dates: First submitted 2010-09-07; First posted 2010-09-09 (Estimated); Last update posted 2010-09-09 (Estimated); Status verified 2010-09

CONDITIONS: Chronic Heart Failure (CHF); Anxiety and Depression; Quality of Life (QOL); Exercise
Keywords: chronic heart failure (CHF); anxiety and depression; quality of life (QOL); exercise
MeSH Terms: conditions — Anxiety Disorders; Depression; Motor Activity; Heart Failure

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Exercise (Experimental)
  Interventions: Other: Home-based exercise

INTERVENTIONS:
Other: Home-based exercise

SUMMARY:
Anxiety and depression are often present in patients with chronic heart failure (CHF). This study aimed to evaluate the influence of anxiety and depression on the physical function, disability, and quality of life (QOL) in CHF. This study examined the effects of 8-week home-based exercise on these parameters, and investigated the correlations between these outcome changes.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of CHF for more than 6 months (NYHA Classes I-III)
* Medically stable for at least 3 months

Exclusion Criteria:

* Malignancy
* Psychiatric disease, primary neuromusculoskeletal or respiratory diseases that affected the assessment of functional or exercise capacity
* Changes in medication occurred during the study period

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2006-12; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Psychologic aspect | 8 weeks
  Anxiety and depression was measured by Hospital Anxiety and Depression Scale (HADS).
Functional capacity | 8 weeks
  Functional capacity was assessed by six-minute walk test (6MWT).
Disability level | 8 weeks
  Groningen Activity Restriction Scale (GARS)
Quality of life | 8 weeks
  Minnesota Living with Heart Failure Questionnaire (MHFQ) was used to assess quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Ying-Tai Wu, Ph.D, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Chien CL, Lee CM, Wu YW, Wu YT. Home-based exercise improves the quality of life and physical function but not the psychological status of people with chronic heart failure: a randomised trial. J Physiother. 2011;57(3):157-63. doi: 10.1016/S1836-9553(11)70036-4. PMID 21843830